CLINICAL TRIAL: NCT04528290
Title: A Phase 1, Randomized, Parallel-group, Open-label, Single-dose, Relative Bioavailability Study of a Pediatric Granule Formulation of Ozanimod in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Relative Bioavailability of a Pediatric Granule Formulation of Ozanimod in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RPC-1063-CP-003; U1111-1256-5078 (Registry Identifier: WHO)
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Healthy Volunteers
Keywords: Ozanimod; RPC-1063; Pediatric Granule Formulation; Healthy Volunteer; Pharmacokinetics (PK)
MeSH Terms: interventions — ozanimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (reference): Current ozanimod capsule formulation (Experimental): Single oral dose of ozanimod 0.92 mg
  Interventions: Drug: Ozanimod
- Group B (test): Ozanimod granule formulation (Experimental): Single oral dose of ozanimod 0.92 mg using Sprinkle capsule. Ozanimod Sprinkle Capsule will be opened, and the entire contents sprinkled onto a teaspoon (5 mL) of applesauce.
  Interventions: Drug: Ozanimod

INTERVENTIONS:
Drug: Ozanimod — Ozanimod capsule formulation of 0.92mg
  Other Names: RPC1063
  Arms: Group A (reference): Current ozanimod capsule formulation
Drug: Ozanimod — Ozanimod, granule formulation of 0.92mg
  Arms: Group B (test): Ozanimod granule formulation

SUMMARY:
This is a Phase 1, open-label, randomized, parallel-group, single-dose study. Approximately 56 participants will be enrolled and randomized into 1 of the 2 treatment groups, with 28 participants in each treatment group as follows:

* Treatment Group A (reference): Current ozanimod capsule formulation
* Treatment Group B (test): Ozanimod granule formulation participants will be screened within 28 days prior to dosing.

Eligible participants will be admitted to the clinical research unit one day before dosing (Day -1) and will be domiciled until Day 15. On Day 1, a single oral dose of 0.92 mg of ozanimod will be administered using either the current capsule formulation (Group A) or the granule formulation (Group B).

Participants will be contacted by telephone 30 ± 5 days after dosing for a follow up safety assessment.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject is a male or female, ≥ 18 and ≤ 55 years
2. Female subjects must meet at least 1 of the following criteria:

   * Negative serum pregnancy test at Screening and Day -1
   * Postmenopausal
   * Received surgical sterilization
3. Female subjects of child-bearing potential:

   Must agree to practice a highly effective method of contraception throughout the study until completion of the Follow-up phone call.

   Highly effective methods of contraception are those that alone or in combination result in a failure rate of a Pearl index of less than 1% per year when used consistently and correctly.

   Acceptable methods of birth control in this study are the following:
   * Combined hormonal (estrogen and progestogen containing) contraception, which may be oral, intravaginal, or transdermal
   * Progestogen-only hormonal contraception associated with inhibition of ovulation, which may be oral, injectable, implantable
   * Placement of an intrauterine device or intrauterine hormone-releasing system
   * Bilateral tubal occlusion
   * Vasectomized partner
   * Complete sexual abstinence

   All subjects:

   Periodic abstinence, withdrawal, spermicides only, and lactational amenorrhea method are not acceptable methods of contraception. Female condom and male condom should not be used together.
4. Subject has a body weight of at least 110 pounds (50 kg); body mass index (BMI) within the range of 18.0 to 30.0 kg/m2
5. Subject is in good health, as determined by no clinically significant findings from medical or surgical history, 12-lead ECG, physical examination, clinical laboratory tests, and vital signs.
6. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
7. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subject with a seated blood pressure outside 90 to 140 mmHg systolic or 50 to 90 mmHg diastolic at Screening or Day -1.
2. Subject with a seated pulse rate outside 55 to 90 beats per minute (bpm) at Screening or Day -1.
3. Subject has a presence or history of any abnormality or illness that, in the opinion of the Investigator, may affect absorption, distribution, metabolism, or elimination of the IPs or would limit the subject's ability to participate in and complete this clinical study.
4. Subject has any condition that confounds the ability to interpret data from the study.
5. Subject has a history of alcoholism, drug abuse, or addiction within 24 months prior to Screening.
6. Subject has a positive serum test for human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV).
7. Subject has used any tobacco- or nicotine-containing products (including but not limited to cigarettes, pipes, cigars, electronic cigarettes, vape, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) or marijuana (cigarette, joint, vape, edibles, etc) within 3 months prior to the first dose of IP.
8. Subject has a positive urine drug test including cotinine at Screening or Day -1.
9. Subject has a positive alcohol urine or breath test at Screening or Day -1.
10. Subject has received any investigational drug within 30 days or 5 times the elimination half-life (if known), whichever is longer, prior to the first dose of IP.
11. Subject has used any systemic over-the-counter medication (excluding acetaminophen up to 1 g/day), dietary or herbal supplement (excluding vitamins/multivitamins) within 7 days prior to the first dose of IP. Herbal supplements including St. John's wort, naringenin, curcurmin/turmeric, passion flower, and quercetin must be discontinued at least 28 days prior to the first dose of IP.
12. Subject has consumed pomelo-variety citrus fruits or juice (including pomelo, grapefruit, Seville oranges) within 7 days prior to the first dose of IP.
13. Subject has used any systemic prescription medication (excluding hormonal contraceptives) within 28 days or 5 times the elimination half-life, whichever is longer, prior to the first dose of IP.
14. Subject has ingested alcohol within 7 days prior to the first dose of IP.
15. Subject fails or is unwilling to abstain from strenuous physical activities for at least 24 hours prior to the first dose of IP.
16. Subject has poor peripheral venous access.
17. Subject has donated greater than 400 mL of blood within 60 days prior to Day 1.
18. Subject with history of any medical condition or medical history that, in the opinion of the Investigator, might confound the results of the study or jeopardize the safety or welfare of the subject.
19. Subject has history of hypersensitivity or allergic reaction to S1P receptor modulators.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic- Cmax (Ozanimod, CC112273, CC1084037) | Up to 14 days
  Maximum observed plasma concentration
Pharmacokinetic- AUC∞(Ozanimod) | Up to 14 days
  Area under the concentration-time curve from time 0 to infinity
Pharmacokinetic- AUClast (CC112273 and CC1084037) | Up to 14 days
  Area under the concentration-time curve from time 0 to last quantifiable concentration

SECONDARY OUTCOMES:
Adverse Events (AEs) | From enrollment until at least 30 days after last dose of IP
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE.
Pharmacokinetic- AUClast (Ozanimod) | Up to 14 days
  Area under the concentration-time curve from time 0 to last quantifiable concentration
Pharmacokinetic- Tmax (Ozanimod, CC112273, and CC1084037) | Up to 14 days
  Time to Cmax
Pharmacokinetic- CL/F (Ozanimod) | Up to 14 days
  Apparent oral clearance
Pharmacokinetic- Vz/F (Ozanimod) | Up to 14 days
  Apparent volume of distribution during terminal phase after oral administration
Pharmacokinetic- t1/2 (Ozanimod, CC112273, and CC1084037) | Up to 14 days
  Terminal elimination half-life

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PPD Phase 1 Clinic, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/